CLINICAL TRIAL: NCT02301611
Title: A Prospective, Randomized, Blinded, Placebo-controlled, Phase IIb Trial of an Autologous Tumor Lysate (TL) + Yeast Cell Wall Particles (YCWP) + Dendritic Cells (DC) Vaccine vs Unloaded YCWP + DC and Embedded Phase I/IIa Trial With Tumor Lysate Particle Only (TLPO) Vaccine in Stage III and Stage IV (Resected) Melanoma to Prevent Recurrence.
Brief Title: Phase IIB TL + YCWP + DC in Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Elios Therapeutics, LLC (Industry)
Collaborators: LumaBridge (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 20141932
Record Dates: First submitted 2014-11-12; First posted 2014-11-26 (Estimated); Results first posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Experimental): autologous TLPLDC (active vaccine)
  Interventions: Drug: TLPLDC
- Placebo (Placebo Comparator): unloaded YCWP + autologous DC (control)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TLPLDC — Autologous tumor lysate, particle-loaded dendritic cell vaccine
  Arms: Treatment
Drug: Placebo
  Arms: Placebo

SUMMARY:
The majority of melanoma vaccines tested to date have been antigen-specific vaccines targeting melanoma-specific or associated antigens and utilizing a variety of delivery systems and immune-adjuvants. As opposed to testing an "off the shelf" vaccine that might be able to treat a subset of patients, our approach has been personalized to the patient and applicable to all patients. Our vaccine approach consists of harnessing the most potent antigen presenting cell in the body - the dendritic cell (DC) - together with the full repertoire of tumor antigens from an individual's cancer. We have conducted phase I and II studies using an autologous DC-tumor cell fusion technique that has now been simplified into a DC-tumor cell lysate vaccine. The autologous tumor lysate (TL) is loaded into yeast cell wall particles (YCWP) that are naturally and efficiently taken up into the patient's DC. These autologous tumor lysate, particle-loaded, DC (TLPLDC) are injected intradermally (ID) monthly x 3 followed by boosters at 6, 12, and 18 months.

DETAILED DESCRIPTION:
Stage III and Stage IV (resected) melanoma patients will be identified prior to definitive surgery and screened for inclusion/exclusion criteria. Eligible patients will be counseled and consented for tissue procurement. Enrolled patients will have their disease surgically resected and a portion 1mg minimum of their melanoma sterilely frozen in provided freezing vials and storage tubes. This tissue will be shipped in liquid nitrogen shippers through FedEx to our central facility in Greenville SC and stored frozen until vaccine preparation. If patients cannot be rendered disease-free, they will be considered screen failures for this study. If melanoma is being resected from multiple locations primary and nodes two different metastatic sites then samples of each would be preferred but not mandatory.

As indicated by SoC per the National Comprehensive Cancer Network (NCCN) guidelines and determined by the treating team, if a patient is to receive systemic therapy (chemotherapy or IFN-aguidelines) and determined by the treating team, if a patient is to receive systemic therapy (chemotherapy or IFN-central facility in Greenville, SC) and stored frozen until vaccine preparation. If patients cannot be rendered disease-free, they will receive a single injection of Neupogen (G-CSF) 300 mod (or its equivalent) SQ 24-48 hrs. prior to having 70 mL of blood collected and sent to our central facility for DC isolation and preparation. Patients who cannot tolerate Neupogen, or its equivalent or refuse it, will have 120 mL of blood drawn and sent. Additional blood may be drawn if additional vaccine doses need to be made or re-made for any reason. Vaccines will be prepared by producing TL through freeze/thaw cycling and then loaded into pre-prepared YCWP. The TL-loaded YCWP will be introduced to the DC for phagocytosis thus creating the TLPLDC vaccine which will be frozen in single dose vials. Each vial will contain 1-1.5 x 106 TLPLDC and will be labeled with the patient's unique study number.

Based on their randomization, autologous TLPLDC (active vaccine) or unloaded YCWP + autologous DC (control) will be sent back to the site in a blinded fashion. Regardless of assigned group, the site will receive 6 single dose vials to be injected intradermal monthly x 3 followed by boosters at 6, 12, and 18 months in the same lymph node draining area (preferably the anterior thigh). Patients must begin vaccinations between 3 weeks and 3 months from completion of (SoC). Frozen tumor will be maintained for active vaccines for all patients to include the control patients. The latter will be offered their active vaccine at time of recurrence in a crossover fashion. Additionally, control patients who do not recur will be offered active vaccine at the completion of the trial.

Safety data will be collected on local and systemic toxicities and graded and reported per the Common Terminology Criteria for Adverse Events (CTCAE) v4.03.

Disease-free status will be monitored per SoC as outlined by NCCN. Suspected recurrences will be documented with biopsy and pathologic confirmation. Time to recurrence will be based on date of randomization to time of confirmed recurrence.

Recurrent patients will be offered participation in the open label portion of the study. New active vaccine will be made for all patients, and they will be inoculated at 0, 1, 2, 3, 6, and 9 mos. Patients will be treated per SoC for their recurrence. Safety and tumor response will be assessed per RECIST and irRC on their SoC follow-up scans.

Blood (50 mL) will be collected from all patients prior to each inoculation and at 24 months from enrollment for a total of 7 time points or a total of 350 mL of blood over 2 years. The collected blood will be sent to our central facility for immunologic testing of the T-cell response.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Eastern Cooperative Oncology Group (ECOG) performance status 0,1 (Appendix D)
* AJCC stage III or IV completely resectable melanoma identified before surgery
* Approximately 1 mg (1 cm3) of accessible and dispensable tumor that will not interfere with pathologic staging
* Clinically disease-free after surgery
* Completing SoC adjuvant therapy per NCCN guidelines to include chemotherapy, radiation therapy, and/or biologic therapy as clinically indicated. (Consent #2 should be signed as close to completion of SoC as possible but may overlap completion by up to one month.)
* Vaccinations initiated between 3 weeks and 3 months from completion of SoC multi-modality cancer care
* Adequate organ function as determined by the following laboratory values:
* ANC ≥ 1,000/μL
* Platelets ≥ 75,000/μL
* Hgb ≥ 9 g/dL
* Creatinine ≤ 1.5 x upper limit of normal (ULN) or Creatinine clearance ≥ 50%
* Total bilirubin ≤ 1.5 ULN
* ALT and AST ≤ 1.5 ULN
* For women of child-bearing potential, agreement to use adequate birth control (abstinence, hysterectomy, bilateral oophorectomy, bilateral tubal ligation, oral contraception, IUD, or use of condoms or diaphragms)
* Signed informed consent

Exclusion Criteria:

* Evidence of residual disease after surgery and SoC adjuvant therapies
* Insufficient tumor available to produce vaccine
* ECOG >2 performance status (Appendix D)
* Immune deficiency disease or known history of HIV, HBV, HCV
* Receiving immunosuppressive therapy including chronic steroids, methotrexate, or other known immunosuppressive agents
* Pregnancy (assessed by urine HCG)
* Breast feeding
* Active pulmonary disease requiring medication to include multiple inhalers (>2 inhalers and one containing steroids)
* Involved in other experimental protocols (except with permission of the other study PI)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2015-01; Primary Completion 2022-05-11 (Actual); Study Completion 2022-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George E Peoples, MD, Study Director — LumaBridge
Locations (18):
- United States (18):
  - University of Alabama Birmingham (UAB) Comprehensive Cancer Center, Birmingham, Alabama
  - Mayo Clinic - Cancer Clinical Research Office, Phoenix, Arizona
  - The University of Arizona Cancer Center, Tucson, Arizona
  - The Angeles Clinic and Research Institute A Cedars-Sinai Affiliate, Los Angeles, California
  - John Wayne Cancer Institute, Santa Monica, California
  - Mount Sinai Cancer Research Program, Miami Beach, Florida
  - Northside Hospital Cancer Institute, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Mayo Clinic, Rochester, Rochester, Minnesota
  - New Mexico Cancer Care Alliance, Albuquerque, New Mexico
  - Laura and Isaac Permutter Cancer Center @ NYU Langone, New York, New York
  - University of Cincinnati Cancer Institute, Cincinnati, Ohio
  - The Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - St. Francis Hospital Cancer Center, Greenville, South Carolina
  - Huntsman Cancer Institute/The University of Utah, Salt Lake City, Utah
  - Providence Regional Medical Center Everett, Everett, Washington

REFERENCES:
- [Derived] Carpenter EL, Van Decar S, Adams AM, O'Shea AE, McCarthy P, Chick RC, Clifton GT, Vreeland T, Valdera FA, Tiwari A, Hale D, Kemp Bohan P, Hickerson A, Smolinsky T, Thomas K, Cindass J, Hyngstrom J, Berger AC, Jakub J, Sussman JJ, Shaheen MF, Yu X, Wagner TE, Faries M, Peoples GE. Prospective, randomized, double-blind phase 2B trial of the TLPO and TLPLDC vaccines to prevent recurrence of resected stage III/IV melanoma: a prespecified 36-month analysis. J Immunother Cancer. 2023 Aug;11(8):e006665. doi: 10.1136/jitc-2023-006665. PMID 37536936
- [Derived] Vreeland TJ, Clifton GT, Hale DF, Chick RC, Hickerson AT, Cindass JL, Adams AM, Bohan PMK, Andtbacka RHI, Berger AC, Jakub JW, Sussman JJ, Terando AM, Wagner T, Peoples GE, Faries MB. A Phase IIb Randomized Controlled Trial of the TLPLDC Vaccine as Adjuvant Therapy After Surgical Resection of Stage III/IV Melanoma: A Primary Analysis. Ann Surg Oncol. 2021 Oct;28(11):6126-6137. doi: 10.1245/s10434-021-09709-1. Epub 2021 Feb 27. PMID 33641012

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients 18 years of age or older with stage III/IV melanoma capable of being disease free after surgery were recruited at the individual study sites. Enrollment start was January 2015. Patients were first randomized 2:1 to receive either the TLPLDC vaccine or placebo (n=124), and then randomization transitioned to 2:1 TLPO or TLPLDC vaccine for 63 more patients. This resulted placebo (n=41), TLPO (n=43), and TLPLDC (n=103) formulations.
Groups:
- Treatment TLPLDC: autologous TLPLDC (active vaccine)
  TLPLDC: Autologous tumor lysate, particle-loaded dendritic cell vaccine
- Placebo: unloaded YCWP + autologous DC (control)
  Placebo
- Treatment TLPO: Tumor Lysate Particle Only (TLPO)
- Treatment TLPLDC-G: autologous TLPLDC - pre-treated with G-CSF
Period: Overall Study
Arm/Group | Treatment TLPLDC | Placebo | Treatment TLPO | Treatment TLPLDC-G
Started | 47 | 41 | 43 | 56
Completed | 19 | 8 | 1 | 8
Not Completed | 28 | 33 | 42 | 48

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment TLPLDC | Placebo | Treatment TLPO | Treatment TLPLDC-G | Total
Number analyzed (Participants) | 47 | 41 | 43 | 56 | 187
Age, Customized [Median (Standard Deviation); unit: years] — Population: Based on stratification
  years
    Age | 69.5 (.07) | 58.7 (.07) | 63.6 (.07) | 61.7 (.07) | 60.2 (.07)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Based on stratification
  Participants
    Female | 16 | 14 | 16 | 16 | 62
    Male | 31 | 27 | 27 | 40 | 125
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Based on stratification
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
    Asian | 0 | 1 | 0 | 0 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 1 | 1 | 0 | 2
    White | 46 | 38 | 41 | 52 | 177
    More than one race | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 1 | 1 | 1 | 3 | 6
Region of Enrollment [Number; unit: participants] — Population: based on stratification factors.
  participants
    United States | 47 | 41 | 43 | 56 | 187

OUTCOME MEASURES:

1. Primary Outcome: Disease Free Survival Assessment
Description: The primary outcome measure of the trial is assessing disease free survival (DFS) at 24 months compared between the vaccinated and control groups after the final enrolled patient completes two years of follow-up. An interim analysis will be performed six months after the final patient is enrolled. This analysis will compare median DFS between vaccinated and control groups.
Time Frame: 24 months
Population: Number of participants remaining at displayed timepoints
Measure: Count of Participants; unit: Participants
Groups:
- Treatment TLPLDC: autologous TLPLDC (active vaccine) Survival Table - remaining cases
Arm/Group | Treatment TLPLDC | Placebo | Treatment TLPO | Treatment TLPLDC-G
Number analyzed (Participants) | 47 | 41 | 43 | 56
Participants
  Survival 6 months | 32 | 30 | 31 | 30
  Survival 12 months | 26 | 20 | 29 | 20
  Survival 18 months | 23 | 12 | 20 | 17
  Survival 24 months | 19 | 7 | 10 | 9

ADVERSE EVENTS:
Time Frame: 36 months
Arm/Group | Treatment TLPLDC | Placebo | Treatment TLPO | Treatment TLPLDC-G
All-Cause Mortality (participants affected / at risk) | 14/47 | 6/41 | 6/43 | 1/56
Serious Adverse Events (participants affected / at risk) | 4/47 | 6/41 | 7/43 | 6/56
Other Adverse Events (participants affected / at risk) | 24/47 | 14/41 | 15/43 | 13/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment TLPLDC (N=47) | Placebo (N=41) | Treatment TLPO (N=43) | Treatment TLPLDC-G (N=56)
Sepsis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Congestive heart failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight loss (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacteremia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Norovirus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Protein calorie malnutrition (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Transient ischemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depressed level of conciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral edema (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment TLPLDC (N=47) | Placebo (N=41) | Treatment TLPO (N=43) | Treatment TLPLDC-G (N=56)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Vestibular disorder (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Endocrine disorder (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Fatigue (General disorders) | 0 (0) | 2 (2) | 3 (3) | 4 (10)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (4)
General muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Athralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 6 (8)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Injection site reaction (Skin and subcutaneous tissue disorders) | 10 (29) | 5 (14) | 5 (6) | 7 (17)
Skin induration (Skin and subcutaneous tissue disorders) | 9 (35) | 4 (20) | 2 (4) | 1 (1)
Pain (at injection site) (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 4 (5) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Oral dysesthesia (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremities (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-02-15): https://cdn.clinicaltrials.gov/large-docs/11/NCT02301611/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-15): https://cdn.clinicaltrials.gov/large-docs/11/NCT02301611/SAP_001.pdf